CLINICAL TRIAL: NCT00255892
Title: Intervention Development for Newly Diagnosed Youth With HIV
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Other Study IDs: ATN 055
Record Dates: First submitted 2005-11-16; First posted 2005-11-21 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-02

CONDITIONS: HIV
Keywords: HIV

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Part A - Provider Interviews: The provider interviews will be comprised of participants who are clinical providers, mental health providers, and case managers with at least 1 year of experience working with HIV-positive youth; one from each category from all 15 ATN sites will be targeted for a total of 45 participants.
- Part B - Youth Focus Groups: The focus groups will be comprised of 6-8 participants per group who are between the ages of 16 and 24, diagnosed HIV+ and aware of their HIV diagnosis for between 12-24 months, and receive services at three selected ATN sites or their community partners for a total of 36-48 participants.
  For the purposes of this study, youth who acquired HIV perinatally will be excluded from participation in this study.

SUMMARY:
This study is an exploratory qualitative investigation of the challenges, strengths, and needed areas of support associated with receiving an HIV diagnosis among youth living with HIV. Qualitative interviews will be conducted with health care providers who work with adolescents living with HIV and focus groups will be conducted with adolescents who are living with HIV (ages 16-24). One third of the focus groups will be conducted in Spanish. Findings from this study will be used to create an outline and development plan for a culturally-sensitive and developmentally appropriate intervention (or set of interventions) for youth recently diagnosed with HIV.

DETAILED DESCRIPTION:
Providers will participate in one interview of approximately one-hour duration; these interviews are expected to occur over a 2 month period. Following the completion of the provider interviews, participants will participate in one 2-hour focus group. A total of 6 focus groups (2 at each of the 3 study sites) are anticipated to occur over a 6-8 week period. The complete study duration is expected to take 12 months.

Part A - Provider interviews - 15 clinical providers, 15 mental health providers, 15 case managers (1 provider from each category per ATN site resulting in a total of 45 interviews).

Part B - Focus groups - 36-48 youth living with HIV. It is estimated there will be 6-8 participants per group and we will conduct two groups at each of three different sites (one male specific group and one female specific group) for a total of six focus groups. One third of the focus groups will be conducted in Spanish.

The provider interviews will be comprised of participants who are clinical providers, mental health providers, and case managers with at least 1 year of experience working with HIV+ youth; one from each category will be interviewed from all 15 ATN sites.

The focus groups will be comprised of participants who are between the ages of 16 and 24, diagnosed HIV+ and aware of their HIV diagnosis for between 12-24 months, and receive services at three selected ATN sites or their community partner.

Focus group participants will be balanced to reflect the diversity (i.e., age, pregnant and parenting women, MSM, mono-lingual Spanish-speaking, etc.) of the clinic populations.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed HIV+ and aware of their HIV status for between 12-24 months
* Between the ages of 16-24 (inclusive)
* Gives informed consent for participation

Exclusion Criteria:

* Presence of serious psychiatric symptoms (active hallucinations, thought disorder)
* Visibly distraught (suicidal, homicidal, exhibiting violent behavior)
* Intoxicated or under the influence of alcohol or other substances at the time of study entry
* Acquired HIV through perinatal infection

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The provider interviews will be comprised of participants who are clinical providers, mental health providers, and case managers with at least 1 year of experience working with HIV+ youth; a target number of one from each category will be interviewed from all 15 ATN sites.
  The focus groups will be comprised of participants who are between the ages of 16 and 24, diagnosed HIV+ and aware of their HIV diagnosis for between 12-24 months, and receive services at one of the three selected ATN sites or their community partner.
  Focus group participants will be balanced to reflect the diversity (i.e., age, pregnant and parenting women, men who have sex with men (MSM), mono-lingual Spanish-speaking, etc.) of the clinic populations.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2006-02; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Elicit information from HIV+ youth and their healthcare providers in order to guide the development of a psychosocial intervention | 4 Months
  To elicit information from HIV+ youth and their healthcare providers in order to guide the development of a psychosocial intervention aimed at improving adjustment to HIV diagnosis among adolescents and young adults recently diagnosed with HIV
Develop an outline and development plan for a culturally-sensitive and developmentally appropriate intervention | 4 Months
  To develop an outline and development plan for a culturally-sensitive and developmentally appropriate intervention (or set of interventions) to improve psychosocial adjustment to an HIV diagnosis among adolescent and young adults recently diagnosed with HIV based on the information collected that is described in Objective 1.

CONTACTS AND LOCATIONS:
Overall Officials: Sybil G. Hosek, PhD, Study Chair — John Stroger Jr. Hospital of Cook County
Locations (3):
- United States (2):
  - Stroger Hospital of Cook County, Chicago, Illinois
  - Montefiore Medical Center, New York, New York
- University of Puerto Rico, School of Medicine, San Juan, Puerto Rico

REFERENCES:
- See also: Website for the Adolescent Trials Network for HIV/AIDS Interventions — http://www.atnonline.org